CLINICAL TRIAL: NCT06443359
Title: Hypofractionated Regional Nodal Irradiation in Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Joshua Dilworth, MD, Radiation Oncology, Corewell Health East
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-226
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: lymphedema; hypofractionated; radiation therapy
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1: sentinel lymph node procedure with or without select removal of clipped lymph nodes (Experimental): Group 1: sentinel lymph node procedure with or without select removal of clipped (clinically involved) lymph nodes. Patients who have more than 5 sentinel lymph nodes removed will be stratified into group 2.
  Interventions: Radiation: hypofractionated radiation
- Group 2: axillary lymph node dissection (Experimental): Group 2: axillary lymph node dissection (with or without sentinel lymph node procedure). Patients who have more than 5 sentinel lymph nodes removed will be stratified into group 2.
  Interventions: Radiation: hypofractionated radiation

INTERVENTIONS:
Radiation: hypofractionated radiation — All patients will receive a dose of 42.56 Gy in 16 daily fractions to the whole breast or chest wall and regional lymph nodes. A boost dose of 10 or 12.5 Gy in 4 or 5 daily fractions of 2.5 Gy, respectively, will be administered to either the lumpectomy cavity or mastectomy scar, as appropriate.

SUMMARY:
This is a prospective clinical trial designed to evaluate the efficacy and safety of hypofractionated regional nodal irradiation in breast cancer patients. After enrollment, participants will be stratified into 2 Groups based on the extent of axillary surgery. Participants will complete activities and assessments at baseline, and after completion of treatment at 1-2 weeks, 3 months, 6 months, 1 year, 2 year, and 3 years following completion of treatment.

DETAILED DESCRIPTION:
This is a prospective clinical trial designed to evaluate the efficacy and safety of hypofractionated regional nodal irradiation in breast cancer patients. Participants are stratified into 2 Groups based on the extent of axillary surgery after enrollment.

Group 1: sentinel lymph node procedure with or without select removal of clipped (clinically involved) lymph nodes.

Group 2: axillary lymph node dissection (with or without sentinel lymph node procedure) or patients who have more than 5 sentinel lymph nodes removed will be stratified into group 2.

Participants will complete activities and assessments at baseline, and after completion of treatment at 1-2 weeks, 3 months, 6 months, 1 year, 2 year, and 3 years following completion of treatment. At baseline consultations, history and physical, lymphedema assessment, toxicity assessment, photographs (optional), patient-reported outcome questionnaire and radiation simulation will be completed. Hypofractionated radiation therapy will be completed weekly through the end of treatment with toxicity assessments. At the 1-2 week follow up, toxicity assessment, photographs (optional) and the patient-reported outcome questionnaire will be completed. At the 3 month, 6 month, 1 year, 2 year and 3 year follow-ups a lymphedema assessment, toxicity assessment, photographs (optional), patient-reported outcome questionnaire and follow up examination will be completed.

All patients will receive a dose of 42.56 Gy in 16 daily fractions to the whole breast or chest wall and regional lymph nodes. A boost dose of 10 or 12.5 Gy in 4 or 5 daily fractions of 2.5 Gy, respectively, will be administered to either the lumpectomy cavity or mastectomy scar, as appropriate. Critical organs will be contoured into the treatment planning such as the heart, left anterior descending artery, ipsilateral lung.

Patients may receive neoadjuvant or adjuvant systemic treatment on this trial. In general, the patient should receive systemic treatment according to the current standard of care at the time of enrollment, taking into account the discretion of the treating medical oncologist.

Expected radiation-related acute adverse events (i.e., those experienced within the first 6 months following treatment) are similar to those with conventionally fractionated radiotherapy and include fatigue and tenderness, pruritus, hyperpigmentation, hypopigmentation, dry desquamation, and moist desquamation of the skin. Potential late effects of radiation include arm lymphedema, shoulder stiffness, fibrosis of normal tissue, telangiectasia, hyperpigmentation, or hypopigmentation of the skin, brachial plexopathy, myositis, rib fracture, pneumonitis, second malignancy, or cardiomyopathy. The participants will be monitored for adverse events during radiotherapy and following radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 18 years old
* Life expectancy of >5 years
* ECOG (Zubrod) performance status 0-1
* Histologically confirmed invasive carcinoma of the breast, including ductal, lobular, mammary, medullary, and tubular histologies
* Clinical T stage of cT0, cT1, cT2, or cT3
* Clinical N stage of cN0, cN1, or cN2a
* Clinical M stage of cM0Definitive surgery must be performed (either partial mastectomy or mastectomy without immediate reconstruction) with negative surgical margins (defined as no invasive tumor or DCIS on ink).
* Must have pathologic T stage of pT1, pT2, or pT3, or if receiving neoadjuvant chemotherapy, ypT0, ypTis, ypT1, ypT2, or ypT3
* Pathologic N stage of pN0, pN1, pN2a, or pN3a, or if receiving neoadjuvant chemotherapy, ypN0,ypN1, ypN2, or ypN3a) NOTE: any patient with clinically involved but undissected lymph nodes that would require a radiation boost will not be eligible.
* The radiation oncologist is planning to treat the breast/chest wall and ipsilateral regional lymphatics (including the axillary, supraclavicular, and internal mammary chains)
* Patient is able to understand and willing to sign an IRB approved written informed consent document
* All dosimetric constraints outlined in protocol section 3.5 can be met

Exclusion Criteria:

* Clinical or pathologic T4 disease, including inflammatory breast cancer
* Clinical N stage of cN2b, cN3 disease, pathologic N stage of pN2b, pN3b, or pN3c disease, or if receiving neoadjuvant chemotherapy, ypN2b, ypN3b, or ypN3c disease
* Radiologic evidence of gross residual disease
* History of prior ipsilateral breast cancer (invasive disease or DCIS)
* Active or history of another malignancy within 5 years of registration with the exception of basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the cervix
* Prior history of radiation therapy to the neck, breast, or thorax. Prior radioactive oral iodine is permitted.
* History of active collagen vascular disease including systemic lupus erythematosis, scleroderoma, or dermatomyositis with an elevated CK level
* Pregnancy, active breast feeding, or refusal or inability to use highly effective means of contraception in participants of child-bearing potential.
* The patient is a prisoner.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with chronic arm lymphedema | 3 years post radiation therapy
  Chronic arm lymphedema will be assessed at the 3 year follow up. Determination of chronic lymphedema will be based on measurements of arm circumference prior to radiation simulation and through the 3 year follow up visit. Clinically significant lymphedema is defined as a 10% or greater difference in ipsilateral arm, forearm, or both, compared to the contralateral side.

SECONDARY OUTCOMES:
Number of participants with recurrence of cancer | 3 years post radiation therapy
  Recurrence will be determined based on the physical exam, imaging and routine follow up visits. This includes local recurrence (ipsilateral breast or chest wall tumor recurrence), regional recurrence (regional lymph nodes, including the ipsilateral axilla (levels 1-3), supraclavicular fossa, or internal mammary chain), locoregional recurrence (local or regional recurrence), and distant metastasis ( outside the ipsilateral breast or ipsilateral regional lymph nodes).
Progress-free survival (months) | 3 years
  This is defined as the number of months participants experienced no locoregional recurrence or distant metastasis from completion date of radiation therapy until the date of progression. The date of progression will be defined as the date of initial suspicion for progression by physical exam or imaging studies.
Overall survival (months) | 3 years
  This is defined as the number of months participants survived from completion date of radiation therapy until the date of death. If a participant is alive, the participant censored at the date of last documentation of the patient being alive.
Number acute toxicities | 6 months
  Number of acute toxicities associated with radiation experienced by participants based on the follow-up assessments at 1-2 weeks, 3 months, 6 months following radiation therapy completion
Number of chronic toxicities | 1 year
  Number of chronic toxicities associated with radiation experienced by participants based on the follow-up assessments completed at 2 weeks, 3 months, 6 months and 12 months following radiation therapy
Cosmetic Outcome | 3 years
  This will be assessment for participants with an intact breast at baseline and at each follow up visit using the Harvard Breast Cosmesis scale. This is a 4-point Likert scale (poor - treated breast seriously distorted, Fair - treated breast clearly difference from untreated breast but not seriously distorted, Good - treated breast slightly different from untreated breast, Excellent - treated breast nearly identical to untreated breast). Cosmetic outcome will be assessed at 1-2 weeks, 3 months, 6 months, 1 year, 2 years, 3 years.
Lymphedema requiring intervention | 3 years
  The number of participants who experience lymphedema requiring intervention such as use of a compression sleeve. This will be determined based on completed follow up assessments.
Participant Perception of Quality of Life | 3 years
  Quality of Life will be assessment using the Cancer Therapy - Breast Cancer (FACT-B) questionnaire. Participants will rate 37 statements on a scale of 0-4 (0 - not at all, 1 - a little bit, 2 - somewhat, 3 - quite a bit, 4 - very much). Negatively worded items are recoded so that a higher score indicates a better quality of life for all items. The FACT-B total score is the sum of scores of all five subscales, ranging from 0 (worst quality of life) to 148 (best quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Dilworth, MD, Principal Investigator — Corewell Health East
Locations (3):
- United States (3):
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan